CLINICAL TRIAL: NCT02866409
Title: Efficacy of Dexmedetomidine as an Adjuvant to Local Anesthetic Agent in Scalp Block and Scalp Infiltration to Control Post Craniotomy Pain
Brief Title: Scalp Block Versus Scalp Infiltration With Dexmedetomidine and Local Anesthetic for Post Craniotomy Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NAVNEH SAMAGH (Other)
Collaborators: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Sponsor-Investigator, NAVNEH SAMAGH, senior resident, Post Graduate Institute of Medical Education and Research, Chandigarh
Organization: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: NK/1062/MD/13422-423
Record Dates: First submitted 2016-08-03; First posted 2016-08-15 (Estimated); Last update posted 2016-08-15 (Estimated); Status verified 2016-08

CONDITIONS: Headache
Keywords: dexmedetomidine; nerve block; anesthesia infiltration
MeSH Terms: conditions — Headache | interventions — Dexmedetomidine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Bupivacaine,dexmedetomidine scalp block (Experimental): Bupivacaine (0.25%) and Dexmedetomedine (1 µg/kg). Maximum dose of bupivacaine kept < 2 mg /kg for scalp block
  Interventions: Procedure: scalp block; Drug: Dexmedetomidine; Drug: Bupivacaine
- bupivacaine dexmedetomidine infiltration (Active Comparator): The incision site was infiltrated with 15-20 ml bupivacaine (0.25%) and dexmedetomedine (1 µg/kg). {1/3rd in the muscle and 2/3rd in the subcutaneous tissue}. Maximum dose of bupivacaine kept less than 2 mg /kg.
  Interventions: Procedure: infiltration; Drug: Dexmedetomidine; Drug: Bupivacaine
- bupivacaine infiltration (Active Comparator): The incision site was infiltrated with 15-20 ml of bupivacaine (0.25%). {1/3rd in the muscle and 2/3rd in the subcutaneous tissue}. Maximum dose of bupivacaine kept less than 2 mg /kg.
  Interventions: Procedure: infiltration; Drug: Bupivacaine

INTERVENTIONS:
Procedure: scalp block — In this group following nerves were blocked-
  1. Supra-orbital nerve
  2. Supra-trochlear nerve
  3. Zygomatico-temporal nerve
  4. Auriculo-temporal nerve
  5. Posterior auricular branches of the greater auricular Nerve
  6. The greater, lesser, and third occipital nerves
  Arms: Bupivacaine,dexmedetomidine scalp block
Procedure: infiltration — The incision site was infiltrated with drug. {1/3rd in the muscle and 2/3rd in the subcutaneous tissue}.
  Arms: bupivacaine dexmedetomidine infiltration; bupivacaine infiltration
Drug: Dexmedetomidine — Dexmedetomidine was administered as a dose of 1 µg/kg in 20 ml 0.25% bupivacaine for scalp block or infiltration.
  Other Names: Precedex; Dexdor
  Arms: Bupivacaine,dexmedetomidine scalp block; bupivacaine dexmedetomidine infiltration
Drug: Bupivacaine — 20 ml of Bupivacaine 0.25% was administered to the patients either in the form of scalp block or infiltration
  Other Names: Marcaine; Sensorcaine; Marcain

SUMMARY:
This study has been designed to assess the efficacy of dexmedetomidine as an adjuvant to local anaesthetic agent bupivacaine in scalp nerve block and scalp infiltration to control post craniotomy pain.A third group where patients were administered bupivacaine only infiltration has also been created.

DETAILED DESCRIPTION:
Patients were randomly allocated into three equal groups by computer generated random numbers. For randomization, the simple random allocation rule was followed, wherein the total sample size (n = 150) was randomly divided into three equal groups. In the event of any case has to be excluded because of requirement of postoperative ventilation, altered sensorium or high grade fever in the post-operative period, the same random number code was allocated to the next patient in order to ensure an equal sample size without any modification to the original random number table. The random numbers were then kept in opaque sealed envelopes, numbered sequentially which were opened just before shifting patient inside operation theatre.

The anaesthesiologist who prepared and administered the study drug were not involved in collection of data. The anaesthesiologist who collected the data from the patient in the postoperative period, the operating surgeon and the patient were blinded to the group assigned to the patient.

Pre-operative Assessment:

Pre-operative anaesthetic evaluation was done on the day prior to the surgery. This included a detailed history regarding physical health, any co-morbid illness, current medications, drug allergy and previous anaesthetic experience. The patient was made familiar about the NRS (0-10, with 0 = no pain, 10 = worst pain ever). A written and informed consent was taken. Patients were fasted and premedicated according to the departmental protocol.

Duration of study period-

Study period started after closure of skin incision of the scalp and continued till 48 hours in the postoperative period

Study groups-

Patients were randomly divided into three groups:

Group BI - Bupivacaine infiltration around surgical incision.

Group BDI - Bupivacaine and dexmedetomidine infiltration around surgical incision

Group BDNB- Bupivacaine and dexmedetomidine used in scalp nerve block.

Anaesthesia Technique-

A standard anaesthesia technique according to the departmental protocol was followed in all the patients. Pre-induction monitoring (Datex- Ohmeda S/5 Avance, Madison, WI, USA) consisted of 5-lead electrocardiography, heart rate, automated non-invasive blood pressure, and pulse oximetry. The patients were then be induced with propofol (1-2 mg/kg) or thiopentone (4-6mg/kg) and trachea were intubated with vecuronium 0.1 mg/kg. Anaesthesia was maintained with intravenous (propofol) or inhalational (isoflurane/sevoflurane/desflurane) anaesthetic agent along with nitrous oxide-oxygen mixture (60:40) and intermittent doses of intravenous vecuronium (0.02 mg/kg). Ventilation was maintained at ETCO2 30 to 35mm Hg. Total fresh gas flow rate was kept at 1-2 L/min. A radial artery catheter was inserted for continuous blood pressure monitoring and blood sampling if indicated. Intraoperative analgesia was maintained with intravenous morphine 0.1mg/kg and morphine repeated at a dose of 0.05 mg/kg if duration of surgery was more than 3 hours. Patients were reversed with neostigmine (0.05mg/kg) and glycopyrolate (0.01mg/kg) after administration of study drugs and were extubated once patient started responding to verbal commands and able to generate adequate tidal volume under spontaneous respiration.

Methods of postoperative analgesia- In all the patients, analgesic procedure was done ensuring proper aseptic precaution at the end of the surgery, after closure of skin incision and before putting the dressings over the incision. Patients were reversed from anaesthesia after the administration of study drugs.

Group BI: The incision site was infiltrated with 15-20 ml of bupivacaine (0.25%). {1/3rd in the muscle and 2/3rd in the subcutaneous tissue}. Maximum dose of bupivacaine kept less than 2 mg /kg.

Group BDI: The incision site was infiltrated with 15-20 ml bupivacaine (0.25%) and dexmedetomedine (1 µg/kg). {1/3rd in the muscle and 2/3rd in the subcutaneous tissue}. Maximum dose of bupivacaine kept less than 2 mg /kg.

Group BDNB: Scalp nerve blocks were given with15-20 ml of combination of Bupivacaine (0.25%) and Dexmedetomedine (1 µg/kg). Maximum dose of bupivacaine kept less than 2 mg /kg.

In this group following nerves were blocked-

1. Supra-orbital nerve
2. Supra-trochlear nerve
3. Zygomatico-temporal nerve
4. Auriculo-temporal nerve
5. Posterior auricular branches of the greater auricular Nerve
6. The greater, lesser, and third occipital nerves

Post-operative assessment:

After extubation patients were shifted to the Post anaesthesia care unit (PACU) and assessed for haemodynamic parameters, sedation and any complication at 15 minutes interval till 2hrs and then at 4, 8, 12, 16, 20, 24, 36 and 48 hours. Assessed for cognitive function at 30 min and 60 min.

Patients were followed after discharge for 6 months by telephonic communication at 1, and 3 month interval for presence of chronic pain.

COLLECTION OF DATA-

Preoperative- Age, sex, weight, ASA status, diagnosis, surgery

Intraoperative-

1. Site of incision
2. Duration of surgery
3. Intra-operative analgesia- morphine in mg/kg

Postoperative-

1. Haemodynamic parameters- Heart rate, systolic and diastolic blood pressure, oxygen saturation was recorded at arrival to PACU and every 15 min interval for 2 hours. Then heart rate and systolic and diastolic blood pressure at 4, 8, 12, 16, 20, 24, 36 and 48 hours after surgery.
2. Respiration rate-was recorded at arrival to PACU and every 15 min interval for 2 hours and then at 4, 8, 12, 16, 20, 24, 36 and 48 hours after surgery.
3. Cognitive function- Patients were evaluated for cognitive function 30 minutes after shifting to PACU using a modified self-devised questionnaire of short orientation memory concentration test.

   Whenever the subjects were able to recall and count with minimal mistakes (1 to 3), were regarded as good, with more than 3 mistakes as fair, and if not be able to recall at all, it was regarded as poor. If the cognitive function outcome was poor then same test was repeated at 1 hour after shifting to PACU. If outcome was again poor, then that patient was excluded from the study.
4. Assessment of pain- Postoperative pain was assessed by Numerical rating scale (NRS) where in 0 shows 'no pain' and 10 shows 'worst imaginable excruciating pain'. It was assessed at arrival to PACU and at 0, 0.5, 1, 1.5, 2, 4, 8, 12, 16, 20, 24, 36 and 48 hours after surgery.
5. Pain free period- Time of first rescue analgesic administration from the time of test drug administration was recorded.
6. Postoperatively rescue analgesic- When NRS score was ≥ 4, rescue analgesic paracetamol 1gm was administered intravenously and total rescue analgesic requirement in 24 and 48 hrs were noted.
7. Rescue drugs to maintain haemodynamic stability- Any adverse events like bradycardia (Heart rate ≤ 40), hypotension (SBP < 90 mm of Hg) were recorded and treated by rescue drugs: atropine-15µg/Kg and mephenteramine-3mg/dose respectively. Total amount of rescue drug requirement in 24 and 48 hours were noted.
8. Postoperative sedation- Level of sedation was assessed using Modified Ramsay Sedation Scale.
9. Adverse events-

   1. Respiratory depressions (Respiration rate < 8 breaths/min) was recorded and managed accordingly.
   2. Postoperative nausea and vomiting (PONV) was assessed on a 4-point scale. and was treated with ondansetron 0.15 mg/kg intravenously if score was >2.

ELIGIBILITY:
Inclusion Criteria:

* Neurosurgical patients
* 18-70 years of age
* ASA class I and II
* Patients undergoing elective craniotomy, who were conscious and oriented to time, person and place and able to understand and use Numerical Rating Scale (NRS)

Exclusion Criteria:

* Patient dull and irritable
* GCS <15
* Craniotomy incision extending beyond scalp (the field of the block) e.g. craniofacial surgery
* Patients treated chronically with analgesics or narcotic medications
* Allergy to local anaesthetics or dexmedetomedine
* Patients planned for post-operative mechanical ventilation

Following patients were excluded from the study during collection of data in the postoperative period:-

* Patients developing fever (≥39°C) in the postoperative period
* Requiring postoperative ventilation (unplanned)
* Having poor cognitive function at 1 hour postoperative period
* GCS <15 in post-operative period.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2013-11; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
post craniotomy pain by Numerical rating scale (NRS) | Immediately after extubation
  Numerical rating scale (NRS) is a scale from 0 to 10 where 0 shows 'no pain' and 10 shows 'worst imaginable excruciating pain
post craniotomy pain by Numerical rating scale (NRS) | 30 minutes after extubation
post craniotomy pain by Numerical rating scale (NRS) | 1 hour after extubation
post craniotomy pain by Numerical rating scale (NRS) | 1.5 hours after extubation
post craniotomy pain by Numerical rating scale (NRS) | 2 hours after extubation
post craniotomy pain by Numerical rating scale (NRS) | 4 hours post extubation
post craniotomy pain by Numerical rating scale (NRS) | 8 hours post extubation
post craniotomy pain by Numerical rating scale (NRS) | 12 hours post extubation
post craniotomy pain by Numerical rating scale (NRS) | 16 hours post extubation
post craniotomy pain by Numerical rating scale (NRS) | 20 hours post extubation
post craniotomy pain by Numerical rating scale (NRS) | 24 hours post extubation
post craniotomy pain by Numerical rating scale (NRS) | 36 hours post extubation
post craniotomy pain by Numerical rating scale (NRS) | 48 hours post extubation

SECONDARY OUTCOMES:
chronic pain using Numerical rating scale (NRS) | 1 month
  Numerical rating scale (NRS) is a scale from 0 to 10 where 0 shows 'no pain' and 10 shows 'worst imaginable excruciating pain
chronic pain using Numerical rating scale (NRS) | 3 months
post operative sedation using Modified Ramsay Sedation Scale | 15 minutes interval till 2hrs post extubation and then at 4, 8, 12, 16, 20, 24, 36 and 48 hours.
  Sedation Score-- by Modified Ramsay Sedation Scale
  1. Anxious/ Agitated/ Restless
  2. Cooperative/ Oriented/ Tranquil
  3. Responds to verbal commands
  4. Brisk response to light glabellar tap or loud noise
  5. Sluggish response to light glabellar tap or loud noise
  6. No Response
post operative sedation using Modified Ramsay Sedation Scale | 4 hours
  Sedation Score-- by Modified Ramsay Sedation Scale
  1. Anxious/ Agitated/ Restless
  2. Cooperative/ Oriented/ Tranquil
  3. Responds to verbal commands
  4. Brisk response to light glabellar tap or loud noise
  5. Sluggish response to light glabellar tap or loud noise
  6. No Response
post operative sedation using Modified Ramsay Sedation Scale | 8 hours.
  Sedation Score-- by Modified Ramsay Sedation Scale
  1. Anxious/ Agitated/ Restless
  2. Cooperative/ Oriented/ Tranquil
  3. Responds to verbal commands
  4. Brisk response to light glabellar tap or loud noise
  5. Sluggish response to light glabellar tap or loud noise
  6. No Response
post operative sedation using Modified Ramsay Sedation Scale | 12 hours.
  Sedation Score-- by Modified Ramsay Sedation Scale
  1. Anxious/ Agitated/ Restless
  2. Cooperative/ Oriented/ Tranquil
  3. Responds to verbal commands
  4. Brisk response to light glabellar tap or loud noise
  5. Sluggish response to light glabellar tap or loud noise
  6. No Response
post operative sedation using Modified Ramsay Sedation Scale | 16 hours.
  Sedation Score-- by Modified Ramsay Sedation Scale
  1. Anxious/ Agitated/ Restless
  2. Cooperative/ Oriented/ Tranquil
  3. Responds to verbal commands
  4. Brisk response to light glabellar tap or loud noise
  5. Sluggish response to light glabellar tap or loud noise
  6. No Response
post operative sedation using Modified Ramsay Sedation Scale | 20 hours.
  Sedation Score-- by Modified Ramsay Sedation Scale
  1. Anxious/ Agitated/ Restless
  2. Cooperative/ Oriented/ Tranquil
  3. Responds to verbal commands
  4. Brisk response to light glabellar tap or loud noise
  5. Sluggish response to light glabellar tap or loud noise
  6. No Response
post operative sedation using Modified Ramsay Sedation Scale | 24 hours.
  Sedation Score-- by Modified Ramsay Sedation Scale
  1. Anxious/ Agitated/ Restless
  2. Cooperative/ Oriented/ Tranquil
  3. Responds to verbal commands
  4. Brisk response to light glabellar tap or loud noise
  5. Sluggish response to light glabellar tap or loud noise
  6. No Response
post operative sedation using Modified Ramsay Sedation Scale | 36 hours.
  Sedation Score-- by Modified Ramsay Sedation Scale
  1. Anxious/ Agitated/ Restless
  2. Cooperative/ Oriented/ Tranquil
  3. Responds to verbal commands
  4. Brisk response to light glabellar tap or loud noise
  5. Sluggish response to light glabellar tap or loud noise
  6. No Response
post operative sedation using Modified Ramsay Sedation Scale | 48 hours.
  Sedation Score-- by Modified Ramsay Sedation Scale
  1. Anxious/ Agitated/ Restless
  2. Cooperative/ Oriented/ Tranquil
  3. Responds to verbal commands
  4. Brisk response to light glabellar tap or loud noise
  5. Sluggish response to light glabellar tap or loud noise
  6. No Response
rescue analgesic requirement in grams | 24 hrs
  total rescue analgesic requirement in grams of paracetamol consumed in 24 hours
rescue analgesic requirement in grams | 48 hrs
  total rescue analgesic requirement in grams of paracetamol consumed in 48 hours

OTHER OUTCOMES:
heart rate in beats per minute(bpm) | 15 minutes interval till 2hrs
  15 minutes interval till 2hrs post extubation
heart rate in beats per minute(bpm) | 4 hours.
heart rate in beats per minute(bpm) | 8 hours.
heart rate in beats per minute(bpm) | 12 hours.
heart rate in beats per minute(bpm) | 16 hours.
heart rate in beats per minute(bpm) | 20 hours.
heart rate in beats per minute(bpm) | 24 hours.
heart rate in beats per minute(bpm) | 36 hours.
heart rate in beats per minute(bpm) | 48 hours.
systolic blood pressure in mm of Hg | 15 minutes interval till 2hrs
  15 minutes interval till 2hrs post extubation
systolic blood pressure in mm of Hg | 4 hours.
systolic blood pressure in mm of Hg | 8 hours.
systolic blood pressure in mm of Hg | 12 hours.
systolic blood pressure in mm of Hg | 16 hours.
systolic blood pressure in mm of Hg | 20 hours.
systolic blood pressure in mm of Hg | 24 hours.
systolic blood pressure in mm of Hg | 36 hours.
systolic blood pressure in mm of Hg | 48 hours.
Diastolic blood pressure in mm of Hg | 15 minutes interval till 2hrs
  15 minutes interval till 2hrs post extubation
Diastolic blood pressure in mm of Hg | 4 hours.
Diastolic blood pressure in mm of Hg | 8 hours.
Diastolic blood pressure in mm of Hg | 12 hours.
Diastolic blood pressure in mm of Hg | 16 hours.
Diastolic blood pressure in mm of Hg | 20 hours.
Diastolic blood pressure in mm of Hg | 24 hours.
Diastolic blood pressure in mm of Hg | 36 hours.
Diastolic blood pressure in mm of Hg | 48 hours.
SpO2 in percentage | 15 minutes interval till 2hours.
SpO2 in percentage | 4 hours.
SpO2 in percentage | 8 hours.
SpO2 in percentage | 12 hours.
SpO2 in percentage | 16 hours.
SpO2 in percentage | 20 hours.
SpO2 in percentage | 24 hours.
SpO2 in percentage | 36 hours.
SpO2 in percentage | 48 hours.
respiratory rate in breaths per minute | 15 minutes interval till 2hrs
  respiratory rate in breaths per minute at 15 minutes interval till 2hrs in post operative period after extubation
respiratory rate in breaths per minute | 4 hours.
Respiratory rate in breaths per minute | 8 hours.
Respiratory rate in breaths per minute | 12 hours.
Respiratory rate in breaths per minute | 16 hours.
Respiratory rate in breaths per minute | 20 hours.
Respiratory rate in breaths per minute | 24 hours.
Respiratory rate in breaths per minute | 36 hours.
Respiratory rate in breaths per minute | 48 hours.
cognitive function using Modified self-devised questionnaire of short orientation memory concentration | 30 minutes
  Modified self-devised questionnaire of short orientation memory concentration test
  1. What date is it today?
  2. What is the current year?
  3. What is his/her birthday?
  4. Count numbers 1 to 10.
  5. Count reverse numbers from 10 to 1.
cognitive function using Modified self-devised questionnaire of short orientation memory concentration | 60 minutes
  Modified self-devised questionnaire of short orientation memory concentration test
  1. What date is it today?
  2. What is the current year?
  3. What is his/her birthday?
  4. Count numbers 1 to 10.
  5. Count reverse numbers from 10 to 1.
post operative nausea vomiting using Postoperative Nausea and Vomiting Scale | 15 minutes interval till 2hrs
  Postoperative Nausea and Vomiting Scale
  1. No PONV: Absence of any emesis or nausea.
  2. Mild PONV: Patient having only mild nausea / one emetic episode / nausea lasting for less than 10 minutes and where no antiemetic is required.
  3. Moderate PONV: Patient has 1-2 emetic episodes / moderate to severe nausea and antiemetic therapy is required.
  4. Severe PONV: Patient has more than 2 emetic episodes / is nauseated more than twice & more than one antiemetic required.
post operative nausea vomiting using Postoperative Nausea and Vomiting Scale | 4 hours.
  Postoperative Nausea and Vomiting Scale
  1. No PONV: Absence of any emesis or nausea.
  2. Mild PONV: Patient having only mild nausea / one emetic episode / nausea lasting for less than 10 minutes and where no antiemetic is required.
  3. Moderate PONV: Patient has 1-2 emetic episodes / moderate to severe nausea and antiemetic therapy is required.
  4. Severe PONV: Patient has more than 2 emetic episodes / is nauseated more than twice & more than one antiemetic required.
post operative nausea vomiting using Postoperative Nausea and Vomiting Scale | 8 hours.
  Postoperative Nausea and Vomiting Scale
  1. No PONV: Absence of any emesis or nausea.
  2. Mild PONV: Patient having only mild nausea / one emetic episode / nausea lasting for less than 10 minutes and where no antiemetic is required.
  3. Moderate PONV: Patient has 1-2 emetic episodes / moderate to severe nausea and antiemetic therapy is required.
  4. Severe PONV: Patient has more than 2 emetic episodes / is nauseated more than twice & more than one antiemetic required.
post operative nausea vomiting using Postoperative Nausea and Vomiting Scale | 12 hours.
  Postoperative Nausea and Vomiting Scale
  1. No PONV: Absence of any emesis or nausea.
  2. Mild PONV: Patient having only mild nausea / one emetic episode / nausea lasting for less than 10 minutes and where no antiemetic is required.
  3. Moderate PONV: Patient has 1-2 emetic episodes / moderate to severe nausea and antiemetic therapy is required.
  4. Severe PONV: Patient has more than 2 emetic episodes / is nauseated more than twice & more than one antiemetic required.
post operative nausea vomiting using Postoperative Nausea and Vomiting Scale | 16 hours.
  Postoperative Nausea and Vomiting Scale
  1. No PONV: Absence of any emesis or nausea.
  2. Mild PONV: Patient having only mild nausea / one emetic episode / nausea lasting for less than 10 minutes and where no antiemetic is required.
  3. Moderate PONV: Patient has 1-2 emetic episodes / moderate to severe nausea and antiemetic therapy is required.
  4. Severe PONV: Patient has more than 2 emetic episodes / is nauseated more than twice & more than one antiemetic required.
post operative nausea vomiting using Postoperative Nausea and Vomiting Scale | 20 hours.
  Postoperative Nausea and Vomiting Scale
  1. No PONV: Absence of any emesis or nausea.
  2. Mild PONV: Patient having only mild nausea / one emetic episode / nausea lasting for less than 10 minutes and where no antiemetic is required.
  3. Moderate PONV: Patient has 1-2 emetic episodes / moderate to severe nausea and antiemetic therapy is required.
  4. Severe PONV: Patient has more than 2 emetic episodes / is nauseated more than twice & more than one antiemetic required.
post operative nausea vomiting using Postoperative Nausea and Vomiting Scale | 24 hours.
  Postoperative Nausea and Vomiting Scale
  1. No PONV: Absence of any emesis or nausea.
  2. Mild PONV: Patient having only mild nausea / one emetic episode / nausea lasting for less than 10 minutes and where no antiemetic is required.
  3. Moderate PONV: Patient has 1-2 emetic episodes / moderate to severe nausea and antiemetic therapy is required.
  4. Severe PONV: Patient has more than 2 emetic episodes / is nauseated more than twice & more than one antiemetic required.
post operative nausea vomiting using Postoperative Nausea and Vomiting Scale | 36 hours.
  Postoperative Nausea and Vomiting Scale
  1. No PONV: Absence of any emesis or nausea.
  2. Mild PONV: Patient having only mild nausea / one emetic episode / nausea lasting for less than 10 minutes and where no antiemetic is required.
  3. Moderate PONV: Patient has 1-2 emetic episodes / moderate to severe nausea and antiemetic therapy is required.
  4. Severe PONV: Patient has more than 2 emetic episodes / is nauseated more than twice & more than one antiemetic required.
post operative nausea vomiting using Postoperative Nausea and Vomiting Scale | 48 hours.
  Postoperative Nausea and Vomiting Scale
  1. No PONV: Absence of any emesis or nausea.
  2. Mild PONV: Patient having only mild nausea / one emetic episode / nausea lasting for less than 10 minutes and where no antiemetic is required.
  3. Moderate PONV: Patient has 1-2 emetic episodes / moderate to severe nausea and antiemetic therapy is required.
  4. Severe PONV: Patient has more than 2 emetic episodes / is nauseated more than twice & more than one antiemetic required.

IPD SHARING:
Plan to Share IPD: Undecided